CLINICAL TRIAL: NCT03921125
Title: The Accuracy of Pleth Variability Index for Directed Fluid Optimization in Donors in Living Donor Liver Transplantation
Brief Title: Pleth Variability Index for Directed Fluid Optimization in Donors in Living Donor Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amr M Hilal Abdou, Lecturer of Anesthesia and Intensive care, Ain Shams University
Other Study IDs: R 53/2018
Record Dates: First submitted 2019-04-17; First posted 2019-04-19 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Fluid Response
Keywords: Living donors; PVI; PPV; Fluids; Response

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Responders
  Interventions: Device: Massimo for Pleth variability index
- Non responders

INTERVENTIONS:
Device: Massimo for Pleth variability index — To assess fluid response
  Groups: Responders

SUMMARY:
In this Study we are trying to validate the accuracy of Plethogram variability index in predicting fluid responsiveness compared to pulse pressure variation in donors of liver transplantation

DETAILED DESCRIPTION:
The liver transplantation program at Ain Shams University Hospitals relies on related living donors. Extra care during anesthetic management of the donor is warranted because of clear ethical considerations.

This prospective observational study was performed after obtaining approval from the ethical committee of the Ain Shams University FWA R 53/2018. Sample of 40 healthy ASA I or II donors' candidate for right lobe hepatectomy for living donor liver transplantation (LDLT) were included and consent was taken. Conventional form of anesthesia was induced with left radial arterial line inserted for invasive blood pressure monitoring, frequent blood gases and lactate sampling, and measuring the PPV, Right insertion of internal jugular vein line for CVP measurement. Fluid management in the form of ringer acetate 3-5 ml/kg/hr recruitment of the patients (Hypovolemic donors) depends on the presenting signs that led the anesthesiologist to decide if the patient's volume status was hypovolemic and in need for fluid replacement without presence of surgical mechanical compression on the IVC or Liver during dissection phase. These diagnostic criteria for volume assessment were heart rate (HR) more than 100 beats/min, systolic arterial blood pressure (SAP) less than 90 mmHg.

Assessment of Hemodynamics during periods of Hypovolemia After exclusion of any surgical mechanical compression, all enrolled hypovolemic patients had left radial arterial line measuring PPV using Drager Monitor and a pulse oximeter measuring PVI using Device Masimo. This device measures the perfusion index which is the indicator of the amplitude of the signal of PVI, confirmation of the wave signal should be obtained from any finger, fingers should be kept warm before test is done. Hypovolemic patients were given a fluid bolus in the form of ringer acetate 5 ml / Kg over 10 minutes. At the end of volume expansion another recorded PPV and PVI are done. Primary outcome was the correlation between PPV and PVI before and after fluid resuscitation

ELIGIBILITY:
Inclusion Criteria:

* Sample of 40 healthy ASA I or II donors' candidate for right lobe hepatectomy for living donor liver transplantation

Exclusion Criteria:

* Lack of consent

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Sample of 40 healthy ASA I or II donors' candidate for right lobe hepatectomy for living donor liver transplantation
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-09-20 (Estimated); Study Completion 2019-10-20 (Estimated)

PRIMARY OUTCOMES:
Correlation between PPV and PVI before and after fluid resuscitation. | 6 hours
  Assess accuracy of device in fluid response

CONTACTS AND LOCATIONS:
Overall Officials: Amr Hilal abdou, Principal Investigator — Ain shams University, Faculty of medicine
Locations (2):
- Egypt (2):
  - Ain Shams University Hospitals, Cairo
  - Ain shams university hospitals, Cairo

IPD SHARING:
Plan to Share IPD: Yes
Decided to share the IPD
Supporting Information: Study Protocol, SAP